CLINICAL TRIAL: NCT01344629
Title: Bioequivalence of Telmisartan Administrated in Two Different Ways: Both in Telmisartan 80 mg/Amlodipine 5 mg Fixed-dose Combination Tablet and Telmisartan 80 mg Tablet and Amlodipine 5mg Tablet in Concomitant Use in Healthy Male Volunteers. (an Open-label, Randomized, Single-dose, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence Study of Telmisartan Between Telmisartan 80 mg/Amlodipine 5 mg FDC Tablet and Telmisartan 80 mg Tab and Amlodipine 5 mg Tab Concomitant Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1235.28
Record Dates: First submitted 2011-04-26; First posted 2011-04-29 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (2):
- Telmisartan80mg/Amlodipin5mg FDC (Experimental): single-dose, four-period replicated crossover design
  Interventions: Drug: Telmisartan/Amlodipin FDC
- Telmisartan80mgtab + Amlodipin5mg tab (Experimental): single-dose, four-period replicated crossover design
  Interventions: Drug: Telmisartan; Drug: Amlodipin

INTERVENTIONS:
Drug: Telmisartan/Amlodipin FDC — Telmisartan80mg/Amlodipin5mg FDC
  Arms: Telmisartan80mg/Amlodipin5mg FDC
Drug: Telmisartan — Telmisartan 80 mg tablet
  Arms: Telmisartan80mgtab + Amlodipin5mg tab
Drug: Amlodipin — Amlodipin 5mg tablet
  Arms: Telmisartan80mgtab + Amlodipin5mg tab

SUMMARY:
To investigate the bioequivalence of telmisartan administrated in two different ways: both in telmisartan 80 mg/amlodipine 5 mg fixed-dose combination tablets (T) and as telmisartan 80 mg tablet and amlodipine 5 mg tablets (R) in concomitant use

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, body temperature), 12-lead electrocardiograms (ECGs), clinical laboratory tests
2. Age: =20 and =35 years
3. Body weight: =50 kg and =80 kg
4. Body mass index (BMI): =18.0 and =25.0 kg/m2

Exclusion criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings in laboratory test results deviating from normal
5. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test
6. History of surgery of the gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Known hypersensitivity to any component of the formulation (telmisartan and amlodipine), to any other angiotensin receptor blocker, or to any other dihydropyridine calcium channel blocker compound
9. Intake of drugs with a long half-life (=24 hours) within at least 1 month or less than 10 half-lives of the respective drug before drug administration
10. Intake of drugs which might reasonably influence the results of the trial on the basis of the knowledge at the time of protocol preparation within 7 days before drug administration
11. Participation in another trial with an investigational drug within 1 months or less than 10 times of half-lives of the investigational products before drug administration
12. Smoker (=20 cigarettes/day)
13. Alcohol abuse (60 g or more ethanol/day: e.g., 3 middle-sized bottles of beer, 3 gous [equivalent to 540 mL] of sake)
14. Drug abuse
15. Blood donation (more than 100 mL within 4 weeks before drug administration)
16. Excessive physical activities (ex. Marathon etc) within 1 week before drug administration
17. Intake of alcohol within 2 days before drug administration
18. Inability to comply with dietary regimen of the study site
19. Inability to refrain from smoking during trial days

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1235.28.001 Boehringer Ingelheim Investigational Site, Kumamoto, Kumamoto, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: T80/A 5mg FDC tablet, Concomitant use, Concomitant use, T80/A 5mg FDC tablet
- Treatment Sequence B: Concomitant use, T80/A 5mg FDC tablet, T80/A 5mg FDC tablet, Concomitant use
Period: Crossover Period 1
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0
Period: Crossover Period 2
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 32 | 32
Completed | 32 | 31
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Crossover Period 3
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0
Period: Crossover Period 4
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Year] | 24.1 (3.3) | 24.5 (3.8) | 24.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz
Description: Area under the concentration-time curve of Telmisartan in plasma over the time interval from 0 to the time of the last quantifiable data point
Time Frame: Serial pharmacokinetic blood samples collected before drug administration, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours after drug administration
Population: One subject who discontinued the study on period 2 was excluded from Pharmacokinetic data set. Therefore, the number of observed PK parameter were 32+32+31+31=126 in T80/A5 FDC tablet and T80 + A5, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 126 | 126
ng*hour/mL | 1970 (67.9) | 1950 (67.0)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 100.9, 90% CI [97.7 to 104.2]

2. Primary Outcome: Cmax
Description: maximum measured concentration of Telmisartan in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 126 | 126
ng/mL | 471 (88.1) | 484 (81.8)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 97.2, 90% CI [87.2 to 108.3]

3. Secondary Outcome: AUC0-∞
Description: area under the concentration-time curve of Telmisartan in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: One subject who discontinued the study on period 2 was excluded from Pharmacokinetic data set. In analysis only used data which the parameter can be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 110 | 112
ng*hour/mL | 2410 (60.4) | 2300 (62.4)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 101.7, 90% CI [98.3 to 105.2]

4. Secondary Outcome: Tmax
Description: time from dosing to the maximum concentration of Telmisartan in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: hour
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 126 | 126
hour | 0.750 (0.500) [0.500 to 4.00] | 0.750 (0.250) [0.250 to 4.00]
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 110.1, 90% CI [95.8 to 124.4]

5. Secondary Outcome: λz
Description: terminal rate constant of Telmisartan in plasma
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: /hour
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 110 | 112
/hour | 0.0297 (52.5) | 0.0326 (45.1)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 91.4, 90% CI [85.6 to 97.6]

6. Secondary Outcome: t1/2
Description: terminal half-life of Telmisartan in plasma
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 110 | 112
hour | 23.3 (52.5) | 21.3 (45.1)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 109.4, 90% CI [102.4 to 116.8]

7. Secondary Outcome: MRTpo
Description: mean residence time of Telmisartan in the body after oral administration
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | T80/A5 mg FDC Tablet | T80mg Tablet and A5 mg Tablet in Concomitant Use
Number analyzed (Participants) | 110 | 112
hour | 21.8 (56.2) | 19.9 (50.5)
Statistical Analysis 1: Comparison: T80/A5 mg FDC Tablet vs T80mg Tablet and A5 mg Tablet in Concomitant Use; Test type: Non-Inferiority or Equivalence — Bioequivalence between T80/A 5mg FDC tablet and T80mg / A5 mg tablet in concomitant use; ANOVA — No statistical test; Test/Reference Ratio of the mean x 100 = 109.0, 90% CI [101.5 to 117.1]

ADVERSE EVENTS:
Time Frame: From signing the informed consent onwards through the observational phase
Arm/Group | Treatment Sequence A | Treatment Sequence B
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.